CLINICAL TRIAL: NCT02509247
Title: Telemonitoring in CPAP Treatment
Acronym: TeleCPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T200/2013
Record Dates: First submitted 2015-06-10; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; CPAP; telemonitoring; telecare
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring group (Experimental): Patients allocated to the telemonitoring group started with wireless telemonitoring after the titration period, i.e. in the beginning of habituation phase of CPAP treatment.
  Interventions: Device: Telemonitoring
- Usual care group (No Intervention): Patients were followed-up during the habituation phase according to hospital's standard procedure.

INTERVENTIONS:
Device: Telemonitoring — Wireless telemonitoring
  Other Names: Restraxx System (ResMed, Sydney, Australia)
  Arms: Telemonitoring group

SUMMARY:
Wireless telemonitoring was used during the habituation phase of continuous positive airway pressure (CPAP) treatment in obstructive sleep apnoea (OSA) patients. Patients were allocated either to the telemonitoring group (n=50) or the usual care group (n=61). Nursing time, patient satisfaction and treatment efficiency and efficacy were compared between the groups at baseline and after one year treatment the CPAP adherence and treatment efficacy were recorded.

DETAILED DESCRIPTION:
Wireless telemonitoring was used during the habituation phase of continuous positive airway pressure (CPAP) treatment in obstructive sleep apnoea (OSA) patients. Patients were allocated either to the telemonitoring group (n=50) or the usual care group (n=61). Nursing time, patient satisfaction and treatment efficiency and efficacy were compared between the groups at baseline and after one year treatment the CPAP adherence and treatment efficacy were recorded.

This study was part of our regular testing and quality assurance procedure when developing and revising clinical treatment protocol of sleep apnoea patients. When planning remarkable changes in treatment protocol we have to test whether it is feasible and cost-effective to change the protocol. The data was retrospectively collected from hospital records and nurses' notes (nursing time). According to instructions of our hospital, the Ethics Committee approval is not required. The approval of the hospital (Head of the Division of Medicine) for testing the wireless telemonitoring system of CPAP treatment was applied and received (Protocol Record T200/2013, diary number TO5/049/13). Written informed consent was obtained from those patients allocated to the telemonitoring group.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients commencing CPAP therapy for OSA

Exclusion Criteria:

* Patient not able to co-operate

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-08; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Nursing time | 3 months
  Nursing time includes patient's visit at nurse office, phone calls, check-ups of telemonitoring data and completing patient records

SECONDARY OUTCOMES:
CPAP adherence measured with in-built clock counter | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tarja Saaresranta, MD, Phd, Principal Investigator — Hospital District of Southwest Finland
Locations (1):
- Turku University Hospital, Turku, Finland